CLINICAL TRIAL: NCT07152496
Title: Integrated Transcriptome-Microbiome Profiling Reveals Host-Microbe Crosstalk in Biliary Dilatation
Brief Title: Host-Microbe Interactions in Biliary Dilatation
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Principal Investigator, Shuo Jin, Associate Chief Physician, Beijing Tsinghua Chang Gung Hospital
Other Study IDs: 24756-0-01
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Choledochal Cyst
Keywords: molecular mechanism; Biliary Dilatation; microbiome
MeSH Terms: conditions — Choledochal Cyst

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — bile duct tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- This group included BD patients
- This group included healthy control

SUMMARY:
This study is an observational cohort study aimed at continuously enrolling patients with biliary dilatation and healthy controls. It will collect bile duct tissue samples and clinical data from participants across all age groups to establish a comprehensive cohort for biliary dilatation research. Based on this cohort, the study seeks to investigate the molecular mechanisms underlying biliary dilatation development and progression, explore the role of host-microbiome interactions in disease processes, and identify biomarkers associated with complications and malignancy risk, to establish evidence-based strategies for improved diagnosis and treatment of biliary dilatation.

DETAILED DESCRIPTION:
Biliary dilatation (BD) is a complex bile duct disease that affects people differently around the world. In Asia, about 1 in every 1,000 people have this condition. In Europe and America, it is much less common, affecting about 1 in every 50,000 to 150,000 people.

People with biliary dilatation face serious health risks. Up to 80% of patients develop complications such as bile duct inflammation (cholangitis) and bile duct stones. Even more concerning, about 30% of patients may develop cancer, and this risk increases with age. Even after surgery to remove the affected bile ducts, patients still face ongoing risks. About 35% continue to have problems with gallstones and bile duct inflammation. Their risk of developing cancer remains 120 to 200 times higher than healthy people, with cancer rates reaching 14.9%.

Despite these serious risks, researchers do not fully understand why biliary dilatation happens, how it gets worse over time, or why it leads to so many complications and such high cancer risk. Very few studies have looked at this disease at the molecular level. One study that examined genes did not find typical genetic changes. Other small studies looking at gene activity and proteins were limited by having too few patients and no comparison groups, so they could not find clear biological patterns.

Recent research has shown that bacteria and other microorganisms play important roles in many bile duct diseases, including bile duct stones, inflammation, and cancer. Because these microorganisms affect so many bile duct conditions, we believe they may also be important in biliary dilatation.

This study aims to create two groups of participants: people with biliary dilatation of all ages and a control group of healthy people. We will collect bile duct tissue samples from patients who have surgery to remove diseased bile ducts and from healthy donor bile duct tissue that would otherwise be discarded during organ transplant surgeries.

Through studying these tissue samples, our research team will work to understand how biliary dilatation develops and gets worse, why complications happen, and what role bacteria and other microorganisms play in this disease process.

ELIGIBILITY:
Inclusion Criteria:

Patients who have been definitively diagnosed with biliary dilatation and are scheduled for surgical resection (Disease group) Healthy donor bile duct tissues discarded during organ transplantation procedures as part of routine surgical preparation (Control group)

Exclusion Criteria:

Patients with severe systemic diseases that may affect study outcomes (Disease group) Insufficient tissue sample quality or quantity (Disease group) Unavailable or inadequate donor bile duct tissue samples (Control group)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Disease Group: Patients diagnosed with biliary dilatation who are scheduled for surgical resection. These participants represent the primary study population for investigating the molecular mechanisms and microbiome characteristics associated with biliary dilatation.
  Control Group: Healthy donor bile duct tissues that are routinely discarded during organ transplantation surgical procedures. These tissues represent normal bile duct samples that are removed as part of standard surgical preparation but are not used for transplantation, serving as healthy controls for comparison of transcriptome and microbiome profiles.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
molecular mechanisms | At the time of surgery.
  Identification of differentially expressed genes and altered molecular pathways in biliary dilatation through integrated transcriptome analysis of bile duct tissue samples, measured by RNA sequencing and bioinformatics analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Shuo Jin, Principal Investigator, Principal Investigator — Beijing Tsinghua Changgeng Hospital
Locations (1):
- Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No